CLINICAL TRIAL: NCT06509828
Title: Expanded Access Protocol for STOMP-II Patients Who Were Unable to Receive Treatment Subsequent to Adipose Tissue Collection (EAP-STOMP2)
Brief Title: Expanded Access Protocol for STOMP-II Patients Who Were Unable to Receive Treatment Subsequent to Adipose Tissue Collection
Acronym: EAP-STOMP2
Status: Available | Type: Expanded Access
Sponsor: Avobis Bio, LLC (Industry)
Collaborators: Alimentiv Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: EAP-STOMP2
Record Dates: First submitted 2024-07-12; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Perianal Fistula Due to Crohn's Disease
Keywords: Matrix plug; Mesenchymal stem cells; Fistula plug; Refractory; Recurrent; STOMP; Autologous
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Biological: AVB-114 — AVB-114 is a mesenchymal cell substrate system comprised of autologous mesenchymal cells incubated with a 3-dimensional bioabsorbable substrate. The drug substance is expanded, pure mesenchymal stem cells (MSC) which are known to modulate local inflammation and orchestrate tissue healing. By incubating cells with a 3-dimensional bioabsorbable substrate designed for anal fistula geometry, cells are locally delivered into the fistula tract to promote healing.

SUMMARY:
The goal of this Expanded Access Protocol is to provide expanded access of AVB-114 to patients who had their fat tissue collected as part of a clinical trial (STOMP-II), but who were subsequently not treated with AVB-114 because they did not meet all eligibility criteria or the investigational product was not successfully manufactured.

DETAILED DESCRIPTION:
AVB-114 is an autologous investigational product under evaluation in Seeded Cells on Matrix Plug Treating Crohn's Perianal Fistulas (STOMP-II; a prospective, multicenter, randomized, blinded outcome assessment, controlled, add-on therapy phase II study) for the treatment of complex perianal fistulas in subjects with Crohn's disease. EAP-STOMP2 is an expanded access protocol for patients who had adipose tissue collected per the STOMP-II protocol, but who were subsequently unable to receive AVB-114 treatment due to screen failure or product manufacturing issues and thus withdrew from the study. Patients will receive AVB-114 as deemed appropriate by investigator and Avobis Bio.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated ICF.
2. Adipose tissue previously collected per the STOMP-II protocol, but were subsequently unable to receive AVB-114 treatment due to screen failure or product manufacturing issues and thus withdrew.
3. Diagnosed with Crohn's disease and a target perianal fistula with one internal opening and at least one external opening.

Exclusion Criteria:

1. Suffer from any condition or illness that, in the opinion of the Investigator, would compromise patient safety.
2. Pregnant, trying to become pregnant, or are breast feeding. Women of childbearing potential (WCBP) and males who have sexual partners that are WCBP must agree to use an adequate method of contraception while participating in this EAP.
3. Known allergies or hypersensitivity to aminoglycosides.
4. History of clinically significant fat-directed autoimmunity.
5. Active, unresolved infection requiring parenteral antibiotics.
6. Unresolved abscess at time of treatment (if screening Pelvic MRI identifies an abscess, it must be resolved before treatment).
7. Target fistula with any of the following characteristics (note that presence of a second fistula tract that is distinctly separate from the target fistula, or a target fistula with a single internal opening and multiple external openings is not exclusionary):

   1. Target fistula has a branching blind ending sinus tract (no external opening) that investigator assesses to be at elevated risk of abscess formation if treated with AVB-114.
   2. Target fistula is a genito-urinary fistula, including rectovaginal (i.e., fistulae that transverse the vaginal canal).
   3. Any anatomical limitation to successfully securing the fistula plug disk.

Sex: All
Age Groups: Child, Adult, Older Adult